CLINICAL TRIAL: NCT01022177
Title: Influence of Acupuncture to Ocular Microcirculation in Patients With Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Professor L.E. Pillunat, University of Dresden, Department of Ophthalmology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AcuDiab1
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- diabetics (Active Comparator): subjects with HbA1c >7,0 and pathological glucose tolerance testing
  Interventions: Procedure: acupuncture
- healthy (Active Comparator): healthy subjects with HbA1c <7,0 and negative glucose tolerance testing
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — acupuncture of the eye in traditional chinese schematics
  Other Names: acupuncture therapy

SUMMARY:
The purpose of this study is to determine the influence of specific eye acupuncture to the ocular microcirculation in diabetic and healthy subjects.

DETAILED DESCRIPTION:
Diabetes is combined with severe vascular damage at the different stages of the disease, causing reduction in retinal perfusion. Acupuncture is supposed to regulate the perfusion. We propose a study to evaluate the effect of acupuncture to the vascular auto regulation in patient with Diabetes, compared to healthy people without vascular or retinal diseases. The perfusion of the retinal vessel will be examined by Retinal vessel analyzer (RVA), Heidelberg retinal Flowmeter (HRF) and the Ocular blood Flowmeter (OBF) before, during and after standardized specific acupuncture at healthy volunteers and patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* persons over 18 years, men or women, diabetic diagnostics within the last year

Exclusion Criteria:

* medical use of anticoagulative substances, use of dorzolamide, use of immunosuppressive medication
* psychiatrics, epileptics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
retinal perfusion by HRF/OBF/RVA | post acupuncture (one day measurement)

CONTACTS AND LOCATIONS:
Overall Officials: Janek - Haentzschel, Dr., Study Director
Locations (1):
- University Carl Gustav Carus, Dresden, Saxony, Germany